CLINICAL TRIAL: NCT03489304
Title: A 6-week Open-Label Study of Treatment of Insomnia With Zaleplon in HIV Positive Patients With Comorbid Depression
Brief Title: Zaleplon in HIV Patients With Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 819083
Record Dates: First submitted 2018-03-27; First posted 2018-04-05 (Actual); Results first posted 2018-09-18 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-04

CONDITIONS: HIV/AIDS; Clinical Depression
Keywords: Insomnia; Zaleplon
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders | interventions — zaleplon

STUDY DESIGN:
Intervention Model Description: 6-week open-label study evaluating zaleplon for insomnia in HIV positive patients with comorbid depression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zaleplon (Other): Open-label zaleplon 5-10mg daily
  Interventions: Drug: Zaleplon

INTERVENTIONS:
Drug: Zaleplon — non-benzodiazepine hypnotic agent

SUMMARY:
In HIV positive patients with sleep onset insomnia and receiving pharmacologic treatment for comorbid depression, the proposed study aims to evaluate the impact of zaleplon on sleep measures determined by insomnia severity index (ISI) and Epworth sleepiness scale (ESS).

DETAILED DESCRIPTION:
An estimated >50% of HIV positive individuals report insomnia. Insomnia and other sleep disturbances negatively impact outcomes in this population by contributing to metabolic dysfunction, reducing quality of life, and impairing psychosocial functioning. Additionally, in HIV depressed populations, insomnia may hinder remission from clinical depression. To date, there have been no pharmacotherapeutic studies treating insomnia in this population, emphasizing the need to determine whether known hypnotic medications work as effectively in HIV positive patients, including those with comorbid depression. Non-benzodiazepine hypnotics represent an attractive pharmacotherapy for treatment of insomnia in a depressed population, as there are reduced side effects and abuse potential compared to classical benzodiazepines. Consequently, an open-label study evaluating zaleplon for insomnia in HIV positive patients with comorbid depression warrants further study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-65 years with a diagnosis of asymptomatic seropositive HIV
2. Principal diagnosis of Major Depressive Disorder or Dysthymic Disorder in accordance with DSM-IV criteria, and receiving pharmacologic treatment.
3. Subject has obtained some subjective benefit from current antidepressant therapy and is agreeable to remain on the same medication for the course of this study
4. Current symptoms of insomnia as determined by a total score of at least 2 on items 4, 5, and 6 of the HAM-D, and specific complaint of sleep onset insomnia (sleep onset latency of at least 1 hour, 3 or more times per week))
5. Free of sleep medication for at least 2 weeks prior to enrollment (we will not enroll any patients who might require weaning off of sedative hypnotic medications in order to be eligible for the study)
6. Ability to understand the requirements of the study and provide informed consent

Exclusion Criteria:

1. Significant chronic, systemic illness or significant neurologic disorder, including traumatic brain injury
2. Clinically significant history of liver disease
3. Psychiatrically unstable patients in the clinical judgment of the investigator as indicated by current acute suicidality, current homicidal thoughts, or current psychosis
4. Lifetime history of schizophrenia, schizoaffective disorder, or any psychotic illness
5. History of substance abuse or dependence over the past 6 months
6. Currently taking medication to assist with sleep (e.g., Ambien/Zolpidem,Dalmane/Flurazepam, Doral/Quazepam, Halcion/Triazolam, Lunesta/Eszopiclone, Prosom/Estazolam, Restoril/Temazepam, Rozerem/Ramelteon, Sonata/Zaleplon, Melatonin, Unisom, Benadryl).
7. Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-03 (Actual); Primary Completion 2015-02-04 (Actual); Study Completion 2015-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Kayser, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Mood & Anxiety Disorders Research and Treatment Program, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zaleplon
Started | 20
Completed | 16
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Zaleplon
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Severity Index (ISI)
Description: The Insomnia Severity Index is a validated sleep scale that measures clinical insomnia severity. The total score ranges from 0-28 where higher values indicate increased severity of insomnia.
Time Frame: Measure at 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zaleplon
Number analyzed (Participants) | 16
score on a scale | 11 (4.5)

2. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: The Epworth Sleepiness Scale (ESS) is a validated sleep scale that quantifies daytime sleepiness across eight domains. The total score ranges from 0-24 where higher values indicate greater daytime sleepiness.
Time Frame: Measure at 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zaleplon
Number analyzed (Participants) | 16
score on a scale | 6.5 (4.9)

3. Secondary Outcome: Quick Inventory of Depressive Symptomatology (QIDS)
Description: The Quick Inventory of Depressive Symptomatology (QIDS) is a validated mood scale that quantifies depression symptoms. The total score ranges from 0-48, where higher values indicate greater depressive symptoms.
Time Frame: Measure at 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zaleplon
Number analyzed (Participants) | 16
score on a scale | 8.7 (6.3)

ADVERSE EVENTS:
Arm/Group | Zaleplon
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No